CLINICAL TRIAL: NCT02037282
Title: A Phase 1, Open Label, Ascending Dose Cohort Study of the Pharmacokinetics of Anti-Influenza Hyperimmune Intravenous Immunoglobulin in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 140043; 14-I-0043
Record Dates: First submitted 2014-01-14; First posted 2014-01-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-12-02

CONDITIONS: Influenza; Flu
Keywords: HAI Titer; Hemagglutination Inhibition Assays; Immunogenicity; Serum Antibody Response
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Drug: Anti-influenza IVIG

SUMMARY:
Despite currently available antivirals, influenza causes significant morbidity and mortality, with 226,000 excess hospitalizations and 30,000-50,000 deaths each year in the United States alone, and more therapies are needed in the armamentarium of anti-influenza medications including humoral immunity-based agents.

This study will evaluate the pharmacokinetics of an anti-influenza hyperimmune intravenous immunoglobulin. Beginning with a low dose, subjects will receive anti-influenza intravenous immunoglobulin (FLU-IVIG) and evaluated on Study Days 0, 3, 7, 14, and 28. The safety and tolerability is evaluated using symptoms, clinical laboratory tests, and pharmacokinetics. Utilizing serum antibody responses as determined by hemagglutination inhibition (HAI) assays, the dose will be escalated as immunogenicity is established....

DETAILED DESCRIPTION:
Despite currently available antivirals, influenza causes significant morbidity and mortality, with 226,000 excess hospitalizations and 30,000-50,000 deaths each year in the United States alone, and more therapies are needed in the armamentarium of anti-influenza medications including humoral immunity-based agents.

This study will evaluate the pharmacokinetics of an anti-influenza hyperimmune intravenous immunoglobulin. Beginning with a low dose, subjects will receive anti-influenza intravenous immunoglobulin (FLU-IVIG) and evaluated on Study Days 0, 3, 7, 14, and 28. The safety and tolerability is evaluated using symptoms, clinical laboratory tests, and pharmacokinetics. Utilizing serum antibody responses as determined by hemagglutination inhibition (HAI) assays, the dose will be escalated as immunogenicity is established.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years and less than or equal to 50 years
  2. Weight less than or equal to 100 kg
  3. Patients must be willing to forgo the seasonal influenza vaccine for 28 days, and the MMR and varicella vaccines for 3 months post infusion of the study drug
  4. Females who are able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 1 effective form of contraception from the date of the subject s signing of the informed consent form through 28 days after the dose of the study drug

EXCLUSION CRIATERIA:

1. Any chronic medical problem that requires daily oral medications (except Tylenol, oral contraceptives, vitamins, and seasonal allergy medications), or other medical history that in the opinion of the investigator significantly increases the risk associated with IVIG
2. Women who are breast-feeding
3. Positive urine or serum pregnancy test
4. Known sensitivity to IVIG
5. IgA < 7 mg/dL
6. Influenza HAI H1N1 > 1:20
7. Receipt of any vaccination within 30 days prior to study drug administration
8. Pre-existing condition that is associated with an increased risk of thrombosis such as cryoglobulinemia, hyper-triglyceridemia, or monoclonal gammopathies
9. Estimated glomerular filtration rate (GFR) < 60 mL/min at screening, calculated using the MDRD formula
10. Medical conditions for which receipt of up to 750 mL volume may be dangerous to the patient (e.g., decompensated congestive heart failure)
11. Abnormal chemistry panel

    -Defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table

    --Evaluating only total CO2 (bicarbonate), creatinine, alkaline phosphatase, ALT, AST, total bilirubin, and estimated GFR by the MDRD equation
12. Abnormal complete blood count (CBC)

    -Defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table

    --Evaluating only the WBC, hemoglobin, hematocrit, and platelets
13. Positive serology for Hepatitis B surface antigen
14. Positive serology for Hepatitis C
15. Positive serology for HIV-1
16. Prior treatment with any investigational drug therapy within 5 half-lives or 30 days, whichever is longer, prior to study drug administration (i.e., Day 0)
17. Receipt of blood products from 30 days prior to study drug administration (i.e., Day 0) through 28 days after the dose of the study drug
18. Presence of any pre-existing illness that, in the opinion of the investigator, would place the patient at an unreasonably increased risk through participation in this study
19. Patients who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-03; Primary Completion 2014-12-02 (Actual); Study Completion 2014-12-02 (Actual)

PRIMARY OUTCOMES:
HAI titer levels predose, at 1 hr post-infusion, and on Days 3, 7, 14 and 28 | 6 months

SECONDARY OUTCOMES:
Type and frequency of adverse events experienced by subjects receiving anti-influenza IVIG by intravenous administration at escalating dose-levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)

REFERENCES:
- [Background] Kumar A, Zarychanski R, Pinto R, Cook DJ, Marshall J, Lacroix J, Stelfox T, Bagshaw S, Choong K, Lamontagne F, Turgeon AF, Lapinsky S, Ahern SP, Smith O, Siddiqui F, Jouvet P, Khwaja K, McIntyre L, Menon K, Hutchison J, Hornstein D, Joffe A, Lauzier F, Singh J, Karachi T, Wiebe K, Olafson K, Ramsey C, Sharma S, Dodek P, Meade M, Hall R, Fowler RA; Canadian Critical Care Trials Group H1N1 Collaborative. Critically ill patients with 2009 influenza A(H1N1) infection in Canada. JAMA. 2009 Nov 4;302(17):1872-9. doi: 10.1001/jama.2009.1496. Epub 2009 Oct 12. PMID 19822627
- [Background] Perez-Padilla R, de la Rosa-Zamboni D, Ponce de Leon S, Hernandez M, Quinones-Falconi F, Bautista E, Ramirez-Venegas A, Rojas-Serrano J, Ormsby CE, Corrales A, Higuera A, Mondragon E, Cordova-Villalobos JA; INER Working Group on Influenza. Pneumonia and respiratory failure from swine-origin influenza A (H1N1) in Mexico. N Engl J Med. 2009 Aug 13;361(7):680-9. doi: 10.1056/NEJMoa0904252. Epub 2009 Jun 29. PMID 19564631
- [Background] Dwyer DE; INSIGHT Influenza Study Group. Surveillance of illness associated with pandemic (H1N1) 2009 virus infection among adults using a global clinical site network approach: the INSIGHT FLU 002 and FLU 003 studies. Vaccine. 2011 Jul 22;29 Suppl 2(0 2):B56-62. doi: 10.1016/j.vaccine.2011.04.105. PMID 21757105